CLINICAL TRIAL: NCT01627418
Title: Warm Homes for Elder New Zealanders: a Community Trial of People With COPD
Brief Title: Warm Homes for Elder New Zealanders
Acronym: WHEZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Otago (Other)
Collaborators: Health Research Council, New Zealand (Other)
Responsible Party: Principal Investigator, Philippa Howden-Chapman, Professor, University of Otago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HRC08/072AR
Record Dates: First submitted 2011-08-02; First posted 2012-06-25 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; CORD; COAD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Voucher (Experimental): Receive the intervention ("Energy Voucher") the first winter enrolled in the study. The intervention is a electricity voucher and a short pamphlet describing how to work out how much heat the voucher can buy.
  Interventions: Behavioral: Energy Voucher
- Control (Other): Receive the intervention the second winter enrolled in the study (thus "No intervention : control arm"). The intervention is a electricity voucher and a short pamphlet describing how to work out how much heat the voucher can buy.
  Interventions: Behavioral: No intervention : control arm

INTERVENTIONS:
Behavioral: Energy Voucher — Receive the intervention the first winter enrolled in the study. The intervention is a electricity voucher and a short pamphlet describing how to work out how much heat the voucher can buy.
  Arms: Voucher
Behavioral: No intervention : control arm — Do not receive the money or pamphlet in the initial study year
  Arms: Control

SUMMARY:
Aim

The purpose of this study is to evaluate whether fuel subsidies reduce exacerbations of COPD among people aged over 55, and therefore whether providing such subsidies is a cost-beneficial policy initiative.

The Warm Homes for Elder New Zealanders Study enrolled community-dwelling people aged over 55 with moderate or worse COPD. Prior to the study commencing the houses were insulated (if feasible, & the house-owner agreed). Data were collected on the health and energy use of the participants.

The households randomly assigned to the "early" intervention group had a subsidy to their power account their first winter in the study. The subsidy was the intervention and was designed to enable the participants, if they chose to do so, to keep their house warmer during the winter.

DETAILED DESCRIPTION:
Warm Homes for Elder New Zealanders (WHEZ)

Background Although there has been considerable recent work on the prevention, management and causes of Chronic Obstructive Pulmonary Disease (COPD), the contribution of housing has not been well researched. This is despite the socio-economic patterning of COPD (Maori women have the highest rate of COPD that has been recorded for any group of women), and the relationship between socio-economic deprivation and housing conditions.

It is likely that improved heating would reduce exacerbations of COPD as:

* COPD patients with the most advanced disease tend to be older people who often live on a fixed income and may be unable to afford adequate heating
* There is a high excess of winter hospitalisations in COPD patients indicating COPD exacerbations may be triggered by cold conditions.
* About one third of exacerbations of COPD are triggered by respiratory infections.
* The Housing, Insulation and Health Study demonstrated a reduction in self-reported respiratory disease after houses were insulated. Therefore improving the heating in households with a COPD patient may reduce respiratory infections and this in turn would reduce the number and severity of exacerbations.

The percentage of people over 65 in New Zealand will increase from 12% to 22% over the next 25 years. Therefore it will become increasingly important to find cost-effective ways of reducing the morbidity of the older age group. As COPD is a significant cause of morbidity amongst older people, this study investigates a potentially cost effective intervention to reduce both the likelihood of expensive hospital stays and improve the quality of life for older people.

Aim To evaluate whether fuel subsidies reduce exacerbations of COPD among people aged over 55, and therefore whether providing such subsidies is a cost-beneficial policy initiative.

Potential Benefits The potential benefits of the study include reducing the burden of disease. The patients and their caregivers may experience improved quality of life. Hospitals may experience fewer patients requiring treatment during the winter. A cost-benefit analysis will quantify the benefits.

ELIGIBILITY:
Inclusion Criteria:

* Post Bronchodilator FEV1/FVC ratio < Lower Limit of Normal (NHanesIII)
* Post Bronchodilator FEV1 < 80% of the predicted FEV1 (NHanesIII)

OR - In the last three years either went to hospital for their COPD or took antibiotics/steriods for their COPD

Exclusion Criteria:

* Not planning to stay in the same dwelling until the end of the study
* Does not want to take part in research
* Unwilling to answer inclusion questionnaire
* Unable to communicate effectively

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2009-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Moderate or severe exacerbations of COPD during winter for which hospitalisation, systemic corticosteroids and/or antibiotics are required to treat the exacerbation | Four months

SECONDARY OUTCOMES:
Severe exacerbations of COPD during winter for which hospitalisation is required to treat the exacerbation | Four months
Moderate exacerbations of COPD during winter; which will be defined as requiring treatment with systemic corticosteroids and/or antibiotics | Four months
All-cause hospitalisation during winter | Four months
Temperature in the living and bedrooms during winter | Four months
Electricity usage during winter | Four months
Costs to health care system of index participant during winter | Four months
Self-reported quality of life for index participant during winter | Four months
Respiratory health of other people living in household during winter | Four months
Any changes in index participant baseline lung function | course of study ( up to 18 months)
Study withdrawals due to death or greater dependency | course of study (up to 18 months)
Support person burden | course of study (up to 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa L Howden-Chapman, PhD, Principal Investigator — University of Otago
Locations (3):
- New Zealand (3):
  - Wellington / Hutt/ Porirua, Wellington, Wellington Region
  - Christchurch, Christchurch
  - Wanganui / Manawatu, Whanganui

REFERENCES:
- [Derived] Viggers HE, Ingham TR, Chapman RB, Crane J, Currie AB, Davies C, Keall M, Howden-Chapman PL. Impact of a Heating Voucher on Health Outcomes in COPD Patients: A Randomised Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2025 Apr 16;20:1097-1109. doi: 10.2147/COPD.S483194. eCollection 2025. PMID 40260082
- [Derived] Viggers H, Howden-Chapman P, Ingham T, Chapman R, Pene G, Davies C, Currie A, Pierse N, Wilson H, Zhang J, Baker M, Crane J. Warm homes for older people: aims and methods of a randomised community-based trial for people with COPD. BMC Public Health. 2013 Feb 26;13:176. doi: 10.1186/1471-2458-13-176. PMID 23442368